CLINICAL TRIAL: NCT05975151
Title: Efficacy and Safety of Pseudomonas Aeruginosa Followed by Postoperative Intravesical Instillation in Patients With Intermediate and High-risk Non-muscle Invasive Bladder Cancer: a Multi-center, Single-arm Clinical Study
Brief Title: Efficacy and Safety of Pseudomonas Aeruginosa for Intermediate and High-risk Non-muscle Invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bks02
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-03

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; NMIBC; Pseudomonas aeruginosa
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Pseudomonas Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pseudomonas aeruginosa Group (Experimental)
  Interventions: Drug: Pseudomonas aeruginosa

INTERVENTIONS:
Drug: Pseudomonas aeruginosa — A total of 63 subjects with intermediate and high risk NMIBC who were scheduled for transurethral resection of bladder tumor (TURBT) from March 2023 in three centers were enrolled in this study. The enrolled patients received submucosal injection of 1U of Pseudomonas aeruginosa injection and bladder irrigation with chemotherapy drugs (gemcitabine, mitomycin C, epirubicin or pirarubicin) immediately after TURBT. After urine was cleared, a sterile urinary catheter was placed, and 10U of Pseudomonas aeruginosa injection and 40ml of normal saline were injected. The perfusion solution was kept for 1 hour, and the position was changed every 20 minutes. The treatment was given once within 24 hours after operation, then once a week for 12 weeks, and then once a month for 12 months in total. Patients were followed up every 3 months after surgery. The last follow-up was completed in February 2025

SUMMARY:
This is a multicenter, single-arm study to evaluate the efficacy and safety of Pseudomonas aeruginosa the treatment of patients with intermediate and high risk non-muscle invasive bladder cancer. The study continued treatment until the patient could not obtain clinical benefits or had intolerable toxic reactions or the patient withdrew the informed consent, whichever occurred first.

DETAILED DESCRIPTION:
This study used a multicenter open single-arm study design. Study start: March 2023 Study end: March 2024 Multi-center: Three centers were selected to conduct the study to avoid differences in efficacy due to differences in operation among centers. Single-arm study: A total of 63 subjects with intermediate-high risk NMIBC who were scheduled for transurethral resection of bladder tumor (TURBT) from March 2023 in three centers were enrolled in this study. The enrolled patients received submucosal injection of 1U of Pseudomonas aeruginosa injection and bladder irrigation with chemotherapy drugs (gemcitabine, mitomycin C, epirubicin or pirarubicin) immediately after TURBT. After urine was cleared, a sterile urinary catheter was placed, and 10U of Pseudomonas aeruginosa injection and 40ml of normal saline were injected. The perfusion solution was kept for 1 hour, and the position was changed every 20 minutes. The treatment was given once within 24 hours after operation, then once a week for 12 weeks, and then once a month for 12 months in total. Patients were followed up every 3 months after surgery. The last follow-up was completed in February 2025.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18 years old, both male and female;
2. Diagnosed as Intermediate or high risk non-muscle invasive bladder cancer, with previous recurrent pathological diagnosis report and cystoscopy available. Intermediate risk was defined as the presence of one or two of the following: multiple tumors, single tumor larger than 3cm, and/or recurrence (≥1 event in low-risk NMIBC within 1 year after diagnosis). High risk was defined as meeting any one of the following: T1 tumor, G3 tumor, carcinoma in situ (CIS), multiple, recurrent and large (> 3cm) TaG1G2/ low-risk tumor (simultaneous);
3. Not receiving BCG or other immune drug infusion chemotherapy at the same time
4. Informed consent and signed informed consent form by patients and their families;
5. Clear consciousness and able to answer questions independently, Patients were asked to complete the questionnaire by themselves;
6. No history of neurological diseases, severe hematological diseases, and dysfunction of heart, lung, liver, or kidney were observed.

Exclusion criteria:

1. Patients with other genitourinary system tumors or other organ tumors;
2. Patients with muscle invasive bladder urothelial carcinoma (≥T2);
3. Patients receiving chemotherapy, radiotherapy or immunotherapy within the past 4 weeks (excluding immediate postoperative intravesical chemotherapy);
4. Pregnant or lactating women, women of childbearing age who did not use effective contraception, and those who planned to become pregnant during the trial (including the partner of male subjects);
5. Known or suspected intraoperative bladder perforation;
6. Gross hematuria was present before enrollment, and the surgical wound was suspected to be unhealed or damaged urinary mucosa;
7. Patients with cystitis, or previous treatment with other intravesical agents, whose bladder irritation significantly affected the evaluation of the study;
8. Patients who had participated in a clinical trial with other drugs within 3 months before enrollment;
9. Patients with known opioid or alcohol dependence;
10. Patients with any condition considered by the investigators to increase the risk of the subject or interfere with the conduct of the trial;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
recurrence rate | 1 year
  Recurrence rate is determined on the basis of cystoscopy

SECONDARY OUTCOMES:
Disease-free survival | 1 year
  Disease-free survival is defined as the time from the start of study treatment to disease recurrence or death from any cause

OTHER OUTCOMES:
adverse event | 2 year
  Adverse events including lower urinary tract symptoms, fever, and gastrointestinal reactions were evaluated according to laboratory and clinical tests (i.e., hematology and blood chemistry, urinalysis, and vital signs) during the observation period

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Jinan, Shandong, China